CLINICAL TRIAL: NCT03945734
Title: Feasibility of Expressive Helping for Chinese-Speaking Cancer Patients and Survivors
Brief Title: Expressive Helping for Chinese-Speaking Cancer Patients and Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-0612
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2021-03

CONDITIONS: Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expressive Helping (Experimental): Participants complete four 20-minute writing/voice-recording sessions spaced one week apart. During the first week, the instructions will explain that cancer patients and survivors benefit from learning about other cancer survivors' experiences. They are told that the first three weeks of writing/voice-recording (writing/talking about their stress and coping at Week 1, deepest emotions about cancer at Week 2, self-affirmation and benefit finding at Week 3) are exercises designed to help them think about their cancer experiences and to prepare them to write/record the narrative they would share on Week 4. During Week 4, they are asked to write/record a narrative as if they are speaking to another Chinese person with cancer, adding advice and encouragements, and reminded that their writing/recording would be shared with other Chinese American cancer patients and survivors.
  Interventions: Behavioral: Expressive Helping

INTERVENTIONS:
Behavioral: Expressive Helping — Expressive helping harnesses the benefits of helping others (e.g., support giving) through writing or voice-recording. Expressive helping integrates two distinct areas of research showing that writing or speaking about ones' negative experiences and engaging in support giving behaviors can improve psychological well-being.

SUMMARY:
This study examines the feasibility, cultural-sensitivity, and health effects of the expressive helping intervention by conducting a single-arm trial with Chinese-speaking cancer patients and survivors.

DETAILED DESCRIPTION:
This study examines whether expressive helping is feasible and culturally-sensitive for Chinese American cancer patients and survivors. For 20 minutes each week over four weeks, participants choose to write or voice-record their thoughts about cancer by following specific prompts designed to help them process their cancer experiences. During the last week of this reflection exercise, participants write or voice-record an anonymous letter to another Chinese cancer patient by sharing their cancer experience and providing advice and encouragement. Health outcomes are assessed at baseline, 1-month, and 3-month follow-ups. A subset of the participants will be invited to share their experiences with the study through qualitative interviews after the last writing/voice-recording session. This research study provides an opportunity for Chinese American cancer patients and survivors to express their feelings without the fear of burdening others, and give them an opportunity to help others by sharing their cancer experiences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer (any type)
* Of Chinese descent
* Over the age of 18
* Can speaking and read Mandarin Chinese

Exclusion Criteria:

* Completed primary cancer treatment more than five years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants screened | through study completion, an average of 1 year
  The number of participants screened for eligibility will be counted.
Compliance rate | through study completion, an average of 1 year
  Compliance rate is calculated by dividing the number of writing/voice-recording sessions finished by the number of sessions assigned.
Retention rate | through study completion, an average of 1 year
  Retention rate is calculated by dividing the number of participants who began the study by the number of participants who finished the entire study.
Meaningfulness of the study | This will be assessed approximately four weeks after the baseline
  We will ask participants open-ended questions about whether they felt participating in this study was meaningful to them.

SECONDARY OUTCOMES:
Change in quality of life as assessed by the Functional Assessment of Cancer Therapy Scale (FACT). | Baseline; 1-month follow-up; 3-month follow-up
  The Functional Assessment of Cancer Therapy Scale (FACT) is a 27-item measure of health-related quality of life (Cella & Tulsky,1993). This scale assesses contains four different subscales, including physical well-being (7 items), social well-being (7 items), emotional well-being (6 items), and functional well-being (7 items).
Change in depressive symptoms as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D). | Baseline; 1-month follow-up; 3-month follow-up
  The CES-D (Radloff, 1977) is a 20-item measure of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No